CLINICAL TRIAL: NCT03305978
Title: Detection of Pulmonary Nodules: Comparison of Ultra-low-dose Chest CT (Approaching a Two Views Chest X-ray Radiation) and Standard Low Dose CT. A Monocentric, Prospective, Non-randomized, Comparative, Open-label Study With Blind Reading of the Judgment Criteria.
Brief Title: Pulmonary Nodule Detection: Comparison of an Ultra Low Dose vs Standard Scan.
Acronym: npUBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: 38RC17.132
Record Dates: First submitted 2017-09-26; First posted 2017-10-10 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Lung Cancer; Smoking; Radiation Exposure
Keywords: Ultra low dose chest CT; lung cancer screening
MeSH Terms: conditions — Lung Neoplasms; Smoking

STUDY DESIGN:
Intervention Model Description: Major Patient Addressed for Thoracic CT without Injection of Contrast
Who Masked: Outcomes Assessor
Masking Description: blinding evaluation of criteria
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultra low dose chest CT (Experimental)
  Interventions: Device: Ultra low dose chest CT
- Low dose chest CT (Active Comparator)
  Interventions: Device: Low dose chest CT

INTERVENTIONS:
Device: Ultra low dose chest CT — An additional ultra low dose CT row is performed for every subject besides standard diagnostic low dose chest CT.
  Other Names: Revolution CT (GE Healthcare) 442507CN0, equiped with ASIR V
  Arms: Ultra low dose chest CT
Device: Low dose chest CT — standard diagnostic low dose chest CT
  Other Names: Revolution CT (GE Healthcare)
  Arms: Low dose chest CT

SUMMARY:
Lung cancer screening programs are still discussed in Europe today, and one of the concern is radiation due to iterative CT. The aim of this monocentric, prospective, non randomized study is to compare an ultra low dose chest CT (approaching a two views X ray) versus a standard low dose chest CT for ≥4mm lung nodules detection, and secondary for lung nodule characterization and smoking associated findings (emphysema, bronchial abnormalities and coronary calcifications).

DETAILED DESCRIPTION:
An additional Ultra Low Dose CT, approaching 0.2mSv, will be performed in consenting patients referred for non enhanced chest CT in our Revolution CT scanner (GE Healthcare®).The dose delivered with the two acquisitions is still lower than the french diagnostic reference level. Standard CT is interpreted and a report is sent to the referent physician as usual. Then the two acquisitions are read over time by two independent radiologists, blinded over judgment criterias. In case of discordance, an other radiologist will arbitrate. We hope to validate our Ultra low dose chest CT protocol, which is more than 10 times less radiating than a standard low dose CT, as a sensitive tool to detect lung nodules.

ELIGIBILITY:
Inclusion criteria :

1. Patients referred for non enhanced chest CT for following indications :

   * lung nodule search or control
   * nodular abnormality on chest X ray
   * statement of COPD or emphysema
   * asbestos exposure
   * nodule localization before radio frequency ablation
   * assessment of disease extent of an extra thoracic cancer (in case of iodinated intravenous contrast agent contraindication)
   * statement before extrathoracic transplantation (in case of iodinated intravenous contrast agent contraindication)
2. Affiliated with the french social security
3. Who signed consent

Exclusion criteria :

1. Inability to lie down and still during the examination
2. Inability to hold breath more than 5 seconds
3. Pneumonia in the last 3 months
4. Body mass index more than 35kg/m²
5. exclusion period of another interventionnal study
6. referred for articles L1121-5 to L1121-8 of french public health code
7. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Ultra low dose CT lung nodule detection sensibility | 22 months
  Detection rate (%) of ≥4mm lung nodules in ultra low dose chest CT versus standard low dose chest CT

SECONDARY OUTCOMES:
Ultra low dose CT diagnostic performances of lung nodule detection | 22 months
  true positives, false positives, true negatives, false negatives, positive predictive value, negative predictive value, specificity, of ≥4mm lung nodules detection within ultra low dose chest CT versus standard low dose chest CT
Concordance of ≥4mm lung nodules characteristics between ultra low dose and standard low dose chest CT | 22 months
  comparison of size, density, type (true nodule or intrapulmonary ganglion) of ≥4mm lung nodule between ultra low dose and standard low dose chest CT
Ultra low dose CT inter-observer reproducibility | 22 months
  inter observer reproducibility for size, density and type of ≥4mm lung nodule detected in ultra low dose CT
Influence of subjects characteristics, nodule location, and nodule size on detection between ultra low dose and standard low dose chest CT | 22 months
  analysis of subjects characteristics (age, gender, body mass index), ≥4mm nodule location, and ≥4 mm nodule size on detection between ultra low dose and standard low dose chest CT
Concordance of emphysema characteristics between ultra low dose and standard low dose chest CT | 22 months
  comparison of emphysema detection, type (centrilobular, paraseptal, panlobular, bullous) and distribution between ultra low dose and standard low dose chest CT
Concordance of coronary calcification detection and quantification between ultra low dose and standard low dose chest CT | 22 months
  Comparison of Weston scores between ultra low dose and standard low dose chest CT
Concordance of bronchial abnormalities evaluation between ultra low dose and standard low dose chest CT | 22 months
  comparison of detection of bronchial thickening or dilatation between ultra low dose and standard low dose chest CT

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Ferretti, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ludwig M, Chipon E, Cohen J, Reymond E, Medici M, Cole A, Moreau Gaudry A, Ferretti G. Detection of pulmonary nodules: a clinical study protocol to compare ultra-low dose chest CT and standard low-dose CT using ASIR-V. BMJ Open. 2019 Aug 15;9(8):e025661. doi: 10.1136/bmjopen-2018-025661. PMID 31420379